CLINICAL TRIAL: NCT01428908
Title: A Phase III Clinical Trial the Immunogenicity and Safety Study of A Group A, C Polysaccharide Meningococcal and Type b Haemophilus Influenzal Conjugate Vaccine in Infants and Children.
Brief Title: Immunogenicity and Safety of A Group A, C Polysaccharide Meningococcal and Type b Haemophilus Influenzal Conjugate Vaccine in Infants and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Royal (Wuxi) Biological Co., LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT007
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Group A, C Polysaccharide Meningitis; Type b Haemophilus Influenza
Keywords: immunogenicity; safety; group A, C polysaccharide meningitis; type b haemophilus Influenza; conjugate vaccine
MeSH Terms: interventions — HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- children group A (Experimental): 600 children aged 2-5 years old, will be vaccinated on day0
  Interventions: Biological: A+C+hib Conjugate Vaccine; Biological: Placebo
- infants group A (Experimental): 600 infants aged 6-23 months old, will be vaccinated on day0, 28
  Interventions: Biological: A+C+hib Conjugate Vaccine; Biological: Placebo
- children group B (Active Comparator): 600 children aged 2-5 years old, will be vaccinated on day0
  Interventions: Biological: A+C Vaccine; Biological: Hib vaccine
- infants group B (Active Comparator): 600 infants aged 6-23 months old, will be vaccinated on day0, 28
  Interventions: Biological: A+C Vaccine; Biological: Hib vaccine

INTERVENTIONS:
Biological: A+C+hib Conjugate Vaccine — The group A, C polysaccharide meningococcal and type b haemophilus influenzal conjugate vaccine (Wuxi Royal Biological Co., LTD, 20110101) will be administered intramuscularly on one arm, per 0.5ml dose
  Arms: children group A; infants group A
Biological: Placebo — Placebo will be administered intramuscularly on the other arm, per 0.5ml dose
  Arms: children group A; infants group A
Biological: A+C Vaccine — The group A, C polysaccharide meningococcal vaccine (Wuxi Royal Biological Co., LTD, 20101202) will be administered intramuscularly on one arm, per 0.5ml dose
  Arms: children group B; infants group B
Biological: Hib vaccine — The type b haemophilus influenzal vaccine (Sanofi Pasteur Limited) will be administered intramuscularly on the other arm, per 0.5ml dose
  Arms: children group B; infants group B

SUMMARY:
Haemophilus influenzae is an important pathogen which can cause primary infection and respiratory viral infection in infants and leaded to secondary infections. The infection of haemophilus is a major cause of morbidity and mortality in infants and children. At present, the developed conjugant Hib vaccine is proved to be safe and effective. Because Hib vaccine can prevent meningitis, pneumonia, epiglottis inflammation and other serious infection caused by Hib bacteria, the WHO suggested that Hib vaccine should be included in the infant's normal immune programming.

Since the use of meningitis aureus polysaccharide vaccine, incidence of a disease in recent years is declined and maintain to the level of 0.5 per 1/100 thousand. But meningitis aureus polysaccharide vaccine with a relatively poor immune response in the infants under the age of two, and the remaining 60% with a low antibody level and a short duration.

According to the present immunization schedule, to reach the median level of antibody levels there are at least 4 doses in need. So it is meaningful to improving vaccine immunogenicity, to provide high levels of long-term protection and to reduce the number of injections.

After the phase I study which was conducted in August, 2011, the safety profile of this vaccine is proved to be acceptable. The phase III study is aimed to further evaluate the safety and the immunization of the vaccine. The objective of this study is to evaluate the safety of the group A, C polysaccharide meningococcal and type b haemophilus influenzal conjugate vaccine.

ELIGIBILITY:
For the children (aged from 2 to 5 years old)

Inclusion Criteria:

* Healthy subjects aged from 2 to 5 years old of normal intelligence.
* The subjects' guardians are able to understand and sign the informed consent.
* Subjects established as healthy after medical history questioning, physical examination and clinical decision and in accordance with vaccination requirements of the investigational vaccine.
* Subjects who can comply with the requirements of the clinical trial program according to the researcher's views.
* Subjects who have never received group A, C polysaccharide meningococcal vaccine and type b haemophilus Influenzal vaccine.
* Subjects with temperature <37°C on axillary setting.

Exclusion Criteria:

* Subject who has a medical history of Meningitis;
* Subject that has a medical history of any of the following: allergies, seizures, epilepsy, encephalopathy history and so on;
* Subject who is allergic with tetanus toxoid components;
* Subject suffering from thrombocytopenia or other coagulation disorder may lead to contraindication to intramuscular injection;
* Subject who has a history of allergic reactions;
* Any known immunological dysfunction;
* Had received gamma globulin or immune globulin, in the past two weeks
* Subject suffering from congenital malformations, dysgenopathy or serious chronic disease;
* Any acute infections
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

For the infants (aged from 6 to 23 months old)

Inclusion Criteria:

* Healthy subjects aged from 6 months to 23 months old of normal intelligence.
* The subjects' guardians are able to understand and sign the informed consent.
* Subjects established as healthy after medical history questioning, physical examination and clinical decision and in accordance with vaccination requirements of the investigational vaccine.
* Subjects who can comply with the requirements of the clinical trial program according to the researcher's views.
* Subjects who have never received group A, C polysaccharide meningococcal vaccine and type b haemophilus Influenzal vaccine.
* Subjects with temperature<37°C on axillary setting.

Exclusion Criteria for the first vaccination:

* Subject who has a medical history of Meningitis;
* Subject that has a medical history of any of the following: allergies, seizures, epilepsy, encephalopathy history and so on;
* Subject who is allergic with tetanus toxoid components;
* Subject suffering from thrombocytopenia or other coagulation disorder may lead to contraindication to intramuscular injection;
* Subject who has a history of allergic reactions;
* Any known immunological dysfunction;
* Had received gamma globulin or immune globulin, in the past two weeks
* Subject suffering from congenital malformations, dysgenopathy or serious chronic disease;
* Any acute infections
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Exclusion Criteria for the second vaccination:

* Had any Grade 3 or Grade 4 adverse reactions or events occurred since the first vaccination
* Any situation meets the exclusion criteria stated in the exclusion criteria for first dose;
* Any condition the investigator believed may affect the evaluation of the vaccine.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2394 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The seroconversion rate of antibody against group A, C polysaccharide meningitis in children after vaccination | 4 weeks (28±3 days) after the vaccination
  to evaluate the seroconversion rate of antibody against group A, C polysaccharide meningitis in children when measured 4 weeks (28±3 days) after the vaccination
The seroconversion rate of antibody against group A, C polysaccharide meningitis in infants after infant series | 4 weeks (28±3 days) after the infant series (two times, 28 day apart)
  to evaluate the seroconversion rate of antibody against group A, C polysaccharide meningitis in infants when measured 4 weeks (28±3 days) after the infant series (two times, 28 day apart).
The seroconversion rate of antibody against type b haemophilus influenza in children after the vaccination | 4 weeks (28±3 days) after the vaccination
  to evaluate the seroconversion rate of antibody against type b haemophilus Influenza in children when measured 4 weeks (28±3 days) after the vaccination
The seroconversion rate of antibody against type b haemophilus influenza in infants after infant series | 4 weeks (28±3 days) after the infant series (two times, 28 day apart)
  to evaluate the seroconversion rate of antibody against type b haemophilus Influenza in infants when measured 4 weeks (28±3 days) after the infant series (two times, 28 day apart)

SECONDARY OUTCOMES:
Injection-site reactions and systemic events after the vaccination in children | 7 days after the vaccination
  to evaluate the injection-site reactions and systemic events of the investigational vaccines in healthy children for 7 days after the vaccination
Injection-site reactions and systemic events after the first vaccination in infants | 7 days after the first vaccination
  to evaluate the injection-site reactions and systemic events of the investigational vaccines in healthy infants for 7 days after the first vaccination
Injection-site reactions and systemic events after the second vaccination in infants | 7 days after the second vaccination
  to evaluate the injection-site reactions and systemic events of the investigational vaccines in healthy infants for 7 days after the second vaccination
GMT of antibody against group A, C polysaccharide meningitis in children after the vaccination | 4 weeks (28±3 days) after the vaccination
  to evaluate the GMT of antibody against group A, C polysaccharide meningitis in children 4 weeks (28±3 days) after the vaccination
GMT of antibody against group A, C polysaccharide meningitis in infants after the infant series | 4 weeks (28±3 days) after the infant series (two times, 28 day apart)
  to evaluate the GMT of antibody against group A, C polysaccharide meningitis in infants 4 weeks (28±3 days) after the infant series (two times, 28 day apart)
GMT of antibody against type b haemophilus Influenza in serum in children after the vaccination | 4 weeks (28±3 days) after the vaccination
  to evaluate the GMT of antibody against type b haemophilus Influenza in children 4 weeks (28±3 days) after the vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Funing county Center for Disease Control and Prevention, Funing County, Jiangsu, China